CLINICAL TRIAL: NCT01807845
Title: Bioavailability of Vitamin D Encapsulated in Casein Micelles, Compared to Its Bioavailability in a Synthetic Emulsifier Currently Used for Supplementation and Enrichment.
Acronym: VD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: No. 1-Version 1.
Record Dates: First submitted 2013-03-07; First posted 2013-03-08 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Vitamin D Deficiency
Keywords: Casein micelles; vitamin D3 (cholecalciferol); Bioavailability; Nanoencapsulation; Nutrition
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Skimmilk VD will be emulsified using Tween 80 (Active Comparator): Skimmilk enriched with VD wherein the VD will be emulsified using Tween 80;
  Interventions: Dietary Supplement: Skimmilk enriched with VD wherein the VD will be emulsified using Tween 80
- Placebo: un-enriched skimmilk. (Placebo Comparator): Placebo: un-enriched skimmilk.
  Interventions: Dietary Supplement: Placebo: un-enriched skimmilk.
- enriched skimmilk with VD (Active Comparator): enriched skimmilk with VD
  Interventions: Dietary Supplement: enriched skimmilk with VD

INTERVENTIONS:
Dietary Supplement: enriched skimmilk with VD — enriched skimmilk with VD
  Arms: enriched skimmilk with VD
Dietary Supplement: Skimmilk enriched with VD wherein the VD will be emulsified using Tween 80 — Skimmilk enriched with VD wherein the VD will be emulsified using Tween 80
  Arms: Skimmilk VD will be emulsified using Tween 80
Dietary Supplement: Placebo: un-enriched skimmilk. — Placebo: un-enriched skimmilk
  Arms: Placebo: un-enriched skimmilk.

SUMMARY:
Background: Vitamin D3 (VD) is an oil soluble vitamin formed in the skin during exposure to UV light. It is essential for bone and calcium metabolism, insulin reactivity, immune system etc. The dietary sources of VD are scarce, and insufficient. Epidemiological studies link proper VD status with lower risks of bone fracture, hypertension, diabetes, cancer and more. VD deficiency is widespread, mainly due to avoidance of sun exposure due to fear of melanoma. Therefore there is an urgent need to enrich staple foods & beverages with VD, to prevent deficiency.

A novel technology was developed , for nanoencapsulating VD within casein micelles (CM) (natural milk protein nanoparticles). Previously we have found that the bioavailability of VD in CM in 1% fat milk was similar to that in an aqueous dietary supplement based on a synthetic emulsifier- Tween 80- which is sometimes used by the industry to add VD into milk.

The main research question studied in the current project is: how will the bioavailability of VD be affected by its delivery in CM compared to its delivery using Tween 80 in a fat free milk product, like nonfat yogurt.

Hypothesis: The open molecular structure of caseins, which evolved to be easily digestible, may facilitate the bioavailability of VD nanoencapsulated in CM, so that it will not be less than that in Tween 80, which is considered to be good. CM are particularly useful for oil-soluble micronutrient delivery in non-fat products. The most widely consumed nonfat milk product is 0% fat yoghurt, chosen it for this study.

Methods: Yoghurts will be made from 3 milk formulations:

1. Skim milk (0% fat) enriched with 50,000 international units (IU) VD in 150 gr product, in CM.
2. Skim milk with same dosage of VD, emulsified with Tween 80.
3. Placebo: skim milk without added VD. 90 healthy adults, aged 18-65, having passed a medical qualification examination, will be randomly assigned to 3 groups. Following over-night fasting they will each consume a 150 gr yoghurt sample as detailed above, and be requested to fast 2 more hours. Blood will be sampled before yoghurt consumption, and after 1, 7 and 14 days following consumption. Blood-serum level of 25(OH)D (the form of VD used as a status indicator in routine blood tests), by chemiluminescence immunoassay (CMIA).

Expected findings: The bioavailability of VD in CM will not be lower than that in Tween 80, in 0% fat yoghurt.

Significance of the study: With the widespread VD deficiency, decreased fat consumption and rising demand for using only natural ingredients there is great importance in delivery of VD and other fat-soluble micronutrients in protein-based delivery systems, like CM, instead of using synthetic emulsifiers, and it is imperative to assure the bioavailability is not compromised by this dramatic change.

CM solubilize VD and help uniformly distribute it in aqueous products and protect it against heat, oxidation and UV.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers . adults aged 18 - 65

Exclusion Criteria:

Intestinal malabsorption, lactose intolerance, medical illness (e.g. liver disease, kidney disease, or diabetes), hypercalcemia, excessive alcohol use, pregnancy, use of medications known to interfere with vitamin D metabolism e.g. anticonvulsants, barbiturates, or steroids), granulomatous disease, use of vitamin D supplements, potential for significant sun exposure (e.g., travel to a sunny vacation site or use of tanning beds) within the month prior to, or during, the study. -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-05 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Serum 25(OH)D level | 0, 1 day, 7 days, 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam-Health Care Campus, Haifa, Israel